CLINICAL TRIAL: NCT04180202
Title: Comparison Study of EzCVP and CVP
Brief Title: Comparison of Non-invasive Vs. Invasive Hemodynamic Measurements
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to inability of clinical site to enroll sufficient number of subjects
Sponsor: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-014-001
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Non-invasive central venous pressure — Non-invasive method to measure central venous pressure indicator
  Other Names: ezCVP; CVPni

SUMMARY:
Comparison of a non-invasive method of measuring central venous pressure to the conventional modality of invasive central venous pressure.

DETAILED DESCRIPTION:
The conventional method used to measure central venous pressure has limitations since it is an invasive procedure that requires a central venous catheter. To overcome this challenge, a new technology to assess CVP non-invasively using an oscillometric method is being developed. It is called enclosed zone central venous pressure (ezCVP). A comparison study of ezCVP and CVP is needed to determine accuracy and reproducibility.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age over 18 years.
2. Arm circumference is 23 cm to 55 cm
3. Subject will have an existing central venous catheter during their ICU stay
4. Subject or legally authorized representative (LAR) is able to understand the risks and potential benefits of participating in the study and is willing to provide written informed consent
5. Subject or LAR is willing and able to comply with protocol procedures

Exclusion Criteria:

1. Finger and/or upper arm anatomical anomaly or disease that may interfere with attaching a pulse oximeter sensor and/or blood pressure cuff.
2. Pregnant (self-reported)
3. Upper extremity deep venous thrombosis currently being treated
4. Severe skin disease involving the upper arm(s)
5. Study investigator may exclude patients based on clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the El Camino Hospital ICU with central venous catheter.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Non-invasive pressure indicator | 12-72 hours
  Evaluate sensitivity and specificity of ezCVP indication based on the case where CVP is in a 'low range' (0 < CVP < 10 mmHg) or 'high range' (>= 10 mmHg)

SECONDARY OUTCOMES:
Direction of change | 12-72 hours
  Correlate the directionality of ezCVP change to invasive CVP change over time (i.e., increasing, decreasing or remaining stable).
Correlation with invasive CVP | 12-72 hours
  Quantify the agreement between ezCVP (non-invasive) and CVP (invasive)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Edmonds, MD, Principal Investigator — Palo Alto Foundation Medical Group
Locations (1):
- El Camino Hospital, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No
Only summary data of participants will be shared.